CLINICAL TRIAL: NCT05991102
Title: Amplitude Modulated Radiofrequency Electromagnetic Field Treatment Combined With TAS-102 (Lonsurf) and Bevacizumab in Refractory Metastatic Colorectal Cancer
Acronym: Live-RF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Pirus Ghadjar, Prof. Dr., Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Live-RF
Record Dates: First submitted 2023-07-21; First posted 2023-08-14 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Refractory Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TAS-102 and Bevacizumab and radiofrequency electromagnetic field treatment (Experimental): Each treatment cycle with TAS-102 will be 28 days in duration.
  One treatment cycle consists of the following:
  * Days 1: Bevacizumab (5 mg/m2/dose) intravenous.
  * Days 1 through 5: TAS-102 (35 mg/m2/dose) orally 2 times daily with the first dose administered in the morning of Day 1 of each cycle and the last dose administered in the evening of Day 5.
  * Days 6 through 7: Recovery
  * Days 8 through 12: TAS-102 (35 mg/m2/dose) orally 2 times daily with the first dose administered in the morning of Day 8 of each cycle and the last dose administered in the evening of Day 12.
  * Days 13 through 28: Recovery
  * Days 15: Bevacizumab (5 mg/m2/dose) intravenously.
  Radiofrequency electromagnetic field treatment using the EHY-2030 device starts within the first week of systemic therapy 2 times weekly (60 min each) with an interval of at least 48h. A modulated electric field with a carrier radiofrequency 13.56 MHz will be generated.
  Interventions: Device: Radiofrequency electromagnetic field treatment

INTERVENTIONS:
Device: Radiofrequency electromagnetic field treatment — Radiofrequency electromagnetic field treatment using a carrier frequency of 13.56 MHz
  Other Names: mEHT; capacitive hyperthermia; electrohyperthermia

SUMMARY:
Combined chemotherapy and radiofrequency electromagnetic field treatment for patients with liver dominant refractory metastatic colorectal cancer

DETAILED DESCRIPTION:
Charité Universitätsmedizin Berlin is currently the only German University Hospital with an available capacitive radiofrequency electromagnetic field treatment device. While there is only data available regarding the low toxicity profile of radiofrequency electromagnetic field treatment for various regions of the body including the abdomen there is no data available on the combined effect of TAS-102 and Bevacizumab and radiofrequency electromagnetic field treatment. The investigators aim to conduct a feasibility trial and plan to compare the results with data of a prospective trial with a comparable patient population.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to any study procedure
* 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically confirmed colorectal cancer
* Liver metastasis
* Patients received at least two prior regimens of standard chemotherapies and the patient is refractory to or failing these therapies or is unsuitable for the treatment.Standard chemotherapy includes fluoropyrimidine, oxaliplatin, irinotecan,bevacizumab and for patients with KRAS wild-type tumors at least one anti-EGFR monoclonal antibody of cetuximab/panitumumab. Patients with BRAF mutant tumors: BRAF inhibitor, MSI-H patients: Checkpoint-inhibition
* Knowledge of KRAS status (i.e. wild-type or mutant)
* Adequate bone-marrow, liver and renal function:

  1. Hemoglobin value of ≥9.0 g/dL.
  2. Absolute neutrophil count of ≥1,500/mm3
  3. Platelet count ≥100,000/mm3 (IU: ≥100 × 109/L).
  4. Total serum bilirubin of ≤1.5 mg/dL
  5. Aspartate aminotransferase and alanine aminotransferase

     ≤3.0 × upper limit of normal (ULN); if liver function abnormalities are due to underlying Liver metastasis, AST and ALT ≤5 × ULN.
  6. Serum creatinine of ≤1.5 mg/dL.
* Patient is able to take medications orally
* Women of childbearing potential with negative pregnancy test and agreement for adequate birth control if conception is possible

Exclusion Criteria:

* Significant extrahepatic metastasis
* Previous treatment with TAS 102
* Serious illness other than colorectal cancer or serious medical condition:

  1. Other concurrently active malignancies excluding malignancies that are disease free for more than 5 years or carcinoma-in-situ deemed cured by adequate treatment.
  2. Known brain metastasis or leptomeningeal metastasis.
  3. Active infection (ie, body temperature ≥38°C due to infection).
  4. Ascites, pleural effusion or pericardial fluid requiring drainage in last 4 weeks
  5. Intestinal obstruction, pulmonary fibrosis, renal failure, liver failure, or cerebrovascular disorder
  6. Uncontrolled diabetes.
  7. Myocardial infarction within the last 12 months, severe/unstable angina, symptomatic congestive heart failure New York Heart Association (NYHA III/IV)
  8. Gastrointestinal hemorrhage.
  9. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or hepatitis B or C.
  10. Patients with autoimmune disorders or history of organ transplantation who require immunosuppressive therapy.
  11. Psychiatric disease that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results.
* Radiofrequency treatment technically not possible (e.g. larger metal implants)
* Cardiac pacemakers/ICD
* Patient not able for supine positioning (e.g. due to pain)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Through study completion, an average of 3 months
  (≥ partial response)

SECONDARY OUTCOMES:
PFS | Through study completion, an average of 6 months
  Progression-free survival
OS | Through study completion, an average of 1 year
  Overall survival
QoL | During 3 years of trial conduction
  European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30
QoL | During 3 years of trial conduction
  European Organisation for Research and Treatment of Cancer (EORTC) QLQ-LMC21
Anxiety and depression | During 3 years of trial conduction
  Hospital Anxiety and Depression Scale (HADS-D)
Acute and late toxicity | During 3 years of trial conduction
  CTCAE version 5

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided